CLINICAL TRIAL: NCT02615457
Title: Huaier Granule in Treating Women With Triple Negative Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Qifeng Yang, Professor, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HECT001
Record Dates: First submitted 2015-11-17; First posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients taking Huaier Granule for adjuvant treatment after the triple negative breast cancer has been surgically removed. The Huaier Granule (Qidong Gaitianli Medicines Co., Ltd.) should be given orally from the 3rd day after surgery up to 5 years after surgery or until study termination.
  Interventions: Drug: Huaier Granule
- Arm II (No Intervention): Patients not taking Huaier Granule after the triple negative breast cancer has been surgically removed.

INTERVENTIONS:
Drug: Huaier Granule — Huaier Granule was given orally, 20 g tid for 5 years.
  Arms: Arm I

SUMMARY:
RATIONALE:

Huaier (Trametes robiniophila Murr) is a traditional Chinese medicine, which has been widely used in China for many years. The investigators previous study has reported that Huaier could exert great inhibitory effects on breast cancer cells both in vitro and in vivo.

PURPOSE:

To evaluate the efficacy and safety of Huaier Granule in treating women who have triple negative breast cancer that has been surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

Compare the disease-free survival (DFS) and overall survival (OS) of patients with triple negative breast cancer who are randomized to adjuvant Huaier Granule group vs. those randomized to Blank-control group.

OUTLINE:

Patients are randomized to the following one of two treatment groups and are followed annually.

Arm I: Patients taking Huaier Granule for adjuvant treatment after the triple negative breast cancer has been surgically removed.

Arm II: Patients not taking Huaier Granule after the triple negative breast cancer has been surgically removed.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 and ≤ 75 years, female;
* Triple negative breast cancer has been surgically removed;
* The triple negative breast cancer has been confirmed by pathological examination and Immunohistochemistry (IHC);
* Not receiving any preoperative anticancer drugs;
* The liver and kidney function satisfies the following conditions within 3 days after surgery (excluding day 3): aspartate aminotransferase (AST), glutamic-oxalacetic transaminase (ALT) < 2 upper limit of normal (ULN), total bilirubin ≤ 1.5 ULN, serum creatinine < 1.5 ULN;
* Other laboratory tests meet the following requirements within 3 days after surgery (excluding day 3): Hb ≥ 90g/l, platelet count ≥ 100×109/L, absolute neutrophil count > 1.5×109/L;
* The expected survival time ≥ 6 months;
* The subjects volunteer to sign the informed consent.

Exclusion Criteria:

* Patients with stage IV breast cancer;
* Triple negative breast cancer was not surgically removed;
* Non-triple negative breast cancer patients confirmed by pathological examination and Immunohistochemistry (IHC);
* Pregnant or lactating women;
* Those with active bleeding due to various reasons;
* Those with HIV infection or AIDS-associated diseases;
* Those with severe acute and chronic diseases;
* Those with severe diabetes;
* Those with serious infectious diseases;
* Those who can not take drugs by oral route;
* Drug abusers or those with psychological or mental diseases that may interfere with study compliance;
* Conditions that are considered not suitable for this study investigators

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-10; Primary Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | Up to 10 years
  Time from randomization to recurrence, metastasis, appearance of a second primary tumor, or death from any cause, whichever occurs first, assessed up to 10 years.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 10 years
  Time from randomization to death from any cause, assessed up to 10 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital of Shandong University, Ji'nan, Shandong, China

REFERENCES:
- [Background] Wang X, Qi W, Li Y, Zhang N, Dong L, Sun M, Cun J, Zhang Y, Lv S, Yang Q. Huaier Extract Induces Autophagic Cell Death by Inhibiting the mTOR/S6K Pathway in Breast Cancer Cells. PLoS One. 2015 Jul 2;10(7):e0131771. doi: 10.1371/journal.pone.0131771. eCollection 2015. PMID 26134510
- [Background] Song X, Li Y, Zhang H, Yang Q. The anticancer effect of Huaier (Review). Oncol Rep. 2015 Jul;34(1):12-21. doi: 10.3892/or.2015.3950. Epub 2015 May 5. PMID 25955759
- [Background] Kong X, Ding X, Yang Q. Identification of multi-target effects of Huaier aqueous extract via microarray profiling in triple-negative breast cancer cells. Int J Oncol. 2015 May;46(5):2047-56. doi: 10.3892/ijo.2015.2932. Epub 2015 Mar 17. PMID 25826742
- [Background] Wang X, Zhang N, Huo Q, Sun M, Dong L, Zhang Y, Xu G, Yang Q. Huaier aqueous extract inhibits stem-like characteristics of MCF7 breast cancer cells via inactivation of hedgehog pathway. Tumour Biol. 2014 Nov;35(11):10805-13. doi: 10.1007/s13277-014-2390-2. Epub 2014 Jul 31. PMID 25077927
- [Background] Wang X, Zhang N, Huo Q, Sun M, Lv S, Yang Q. Huaier aqueous extract suppresses human breast cancer cell proliferation through inhibition of estrogen receptor alpha signaling. Int J Oncol. 2013 Jul;43(1):321-8. doi: 10.3892/ijo.2013.1947. Epub 2013 May 20. PMID 23686317
- [Background] Wang X, Zhang N, Huo Q, Yang Q. Anti-angiogenic and antitumor activities of Huaier aqueous extract. Oncol Rep. 2012 Oct;28(4):1167-75. doi: 10.3892/or.2012.1961. Epub 2012 Aug 8. PMID 22895629
- [Background] Zhang N, Kong X, Yan S, Yuan C, Yang Q. Huaier aqueous extract inhibits proliferation of breast cancer cells by inducing apoptosis. Cancer Sci. 2010 Nov;101(11):2375-83. doi: 10.1111/j.1349-7006.2010.01680.x. PMID 20718753